CLINICAL TRIAL: NCT01254149
Title: Intraocular Pressure Lowering Effects of Topical Anesthetics Used Frequently in the Ophthalmology Clinic
Brief Title: IOP Lowering Effects of Topical Anesthetics Used Frequently in the Ophthalmology Clinic
Status: Completed | Type: Observational
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Other Study IDs: 0577-10-FB
Record Dates: First submitted 2010-12-02; First posted 2010-12-06 (Estimated); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Normal Tension Glaucoma
MeSH Terms: conditions — Low Tension Glaucoma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The primary purpose of this study is to determine whether topical ophthalmic anesthetics lower the intraocular pressure in the eye.

DETAILED DESCRIPTION:
Each day almost all patients in an ophthalmology clinic get their intraocular pressure of each eye measured. This measurement is used to make important decisions regarding risk of dilation and also is essential in the management of glaucoma patients, as intraocular pressure (IOP) remains one of the only modifiable factors in glaucoma. The intraocular pressure is also measured in an eye that has undergone an operative procedure where pressures can increase to dangerous levels signaling the need for immediate intervention.

In most ophthalmology clinics the intraocular pressure is measured via Goldmann applanation tonometry, which is considered the standard method of measurement. The Goldmann tonometer is a device that uses an applanation prism to flatten a small portion of the cornea to measure the eye. The pressure within the eye is determined by how much force is needed to flatten the cornea. In order to perform the test the subject receives a topical anesthetic and fluorescein sodium dye on the surface of the eye. The intraocular pressure is all frequently measured in ophthalmology by pneumatonometry and the Tonopen. These two additional methods of contact tonometry measure the amount of force needed to displace the cornea and then calculate the intraocular pressure1. Both require instillation of topical anesthetic eye drops prior to measuring the pressure, cut these latter two methods require no dye. The principal anesthetics used in the United States are proparacaine or benoxinate. For Goldmann applanation, these anesthetics must be combined with a fluorescein dye.

Both proparacaine and benoxinate are esters of para-aminobenzoic acid (PABA) that are used for topical ophthalmic anesthesia. Both have onset of action in approximately 10-20 seconds and both duration of action of 10-20 minutes. They provide sufficient anesthesia to permit minor procedures involving the superficial cornea and conjunctiva. Proparacaine is commonly used alone, but can be purchased pre-mixed with fluorescein dye, whereas, benoxinate is only available in combination with fluorescein dye1. Fluorescein sodium is a yellow acid dye from the xanthenes family that absorbs light of the 493 nanometer wavelength (blue) and then emits or fluoresces light of 520 nanometer wavelength (yellow-green). This dye is ubiquitous in ophthalmologic practices as it is used both intravenously and topically to assist in making ophthalmologic diagnoses1.

For contact tonometry, one of these topical anesthetics is traditionally instilled in each eye and the intraocular pressure is then measured. This is typically done by a technician first, and if there is any question regarding the measurement it is repeated again by the physician seeing the patient. In academic institutions the intraocular pressure may also be routinely checked additional times by the resident. For certain patients suspected of having glaucoma the intraocular pressure variation throughout the day is monitored in what is called a diurnal curve measurement. With this test, the intraocular pressure may be checked upwards of ten (10) times in a single day (each measurement with an additional instillation of topical anesthetic). All of these examinations are done with minimal danger and with little discomfort for the patient.

Despite this standard protocol for measurement of the intraocular pressure, it has been suggested that the very anesthetic agents we use to measure the pressure may actually cause some lowering of the intraocular pressure. In rabbits proparacaine has recently been shown to reduce episcleral venous pressure, an important component of the intraocular pressure, and the intraocular pressure itself (Zamora). Attempts to show the pressure lowering effect of these frequently used topical anesthetics in humans using our traditional intraocular measurement devices has been difficult as all three methods mentioned above require topical anesthetic. Some European studies have used non-contact tonometry to verify these findings. For example, Montero et al used non-contact tonometry to determine the effect of the topical anesthetics and found that there was a statistically significant decrease in the intraocular pressure after application of topical anesthetic3. Baudouin et al also found that, when measured via non-contact tonometry, some topical anesthetics lower the intraocular pressure4. In their study the topical anesthetics, oxybuprocaine and betoxycaine used more frequently in the United States. Both of these studies were done using non-contact tonometry. Traditionally with non-contact tonometry, a puff of air is directed towards the corneal surface and the displacement of the corneal surface is measured and used to estimate the intraocular pressure. However, in the United States most ophthalmology offices rely on contact tonometry to evaluate the intraocular pressure rather than non-contact tonometry. Based on our review of the literature, no one has yet measured the intraocular pressure lowering effects of these topical anesthetics with contact tonometry.

There is a currently a device on the market which is approved by the Food and Drug Administration that is able to measure intraocular pressure via contact tonometry that does not require use of topical anesthetic drops. This device is sold as the ICare tonometer. The ICare is a tonometer that uses a rebound technology in which a very light-weight probe is used to make momentary contact with the cornea. In rebound technology, the motion parameters of the probe are recorded during the measurement. An induction based coil system and advanced algorithms analyze the probe deceleration, contact time and other parameters as the probe touches the cornea. The deceleration and rebound parameters change as a function of the intraocular pressure. The tonometer is preprogrammed for six measurements, discarding the highest and lowest intraocular pressure readings, and calculating the average pressure value. The pressure is recorded in millimeters of mercury (mmHg). No anesthesia is involved because the touch of the probe is so gentle that intraocular pressure measurement is barely noticed by the subject5. The ICare is currently used on patients in our clinic for whom the traditional intraocular pressure measurement devices have not been appropriate like newborns and infants. It does not require topical anesthesia and recent data supports that its intraocular pressure measurements are reliable6,7. Thus, the ICare tonometer finally provides a way to use contact tonometry to verify whether or not the two most commonly used topical anesthetics lower intraocular pressure.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be 19 years of age and older

Exclusion Criteria:

* Corneal diseases including corneal transplants, corneal dystrophies, or trauma to the cornea that may prevent reliable tonometry of either eye.
* Intolerant to topical Proparacaine and Benoxinate
* Pregnant or nursing
* 18 years of age and younger.
* Physical limitation preventing ability to obtain reliable intraocular measurements (e.g. difficulty positioning subjects in front of the slit lamp or inability to keep eyes open during the intraocular pressure checks).

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects 19 years of age and older with normal eyes and with ocular disease.
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2011-01-17 (Actual); Primary Completion 2012-04-01 (Actual); Study Completion 2012-04-01 (Actual)

PRIMARY OUTCOMES:
Measured pressures in subjects' eyes with and without anesthetics. | 30 minutes
  Intraocular pressure is measured via Goldmann applanation tonometry, which is considered the standard method of measurement with and without anesthetics.

CONTACTS AND LOCATIONS:
Overall Officials: Nathan Welch, MD, Principal Investigator — UNMC Department of Ophthalmology and Visual Sciences
Locations (1):
- University of Nebraska Medical Center, Department of Ophthalmology, Omaha, Nebraska, United States